CLINICAL TRIAL: NCT02618356
Title: A Phase II Clinical Study of Combined Use of Raltitrexed and S-1 as Treatment for Patients With Metastasizing Colorectal Cancer Failed of Standard Chemotherapy
Brief Title: Combined Use of Raltitrexed and S-1 as Treatment for Patients With Metastasizing Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Weijian Guo, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: guoweijian-2015-RS
Record Dates: First submitted 2015-11-17; First posted 2015-12-01 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Metastatic Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — raltitrexed; S 1 (combination); gimeracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- combined use Raltitrexed and S-1 (Experimental): Raltitrexed 3mg/m2 intravenously guttae, d1 and S-1,bid,po,d1-d14,every three weeks for a cycle.
  BSA(body surface area) S-1 dosage <1.25 m2 80 mg/d
  * 1.25m2 - <1.5 m2 100 mg/d
  * 1.5 m2 120 mg/d
  Interventions: Drug: Raltitrexed and S-1

INTERVENTIONS:
Drug: Raltitrexed and S-1 — Raltitrexed 3mg/m2 intravenously guttae, d1 and S-1,bid,po,d1-d14,every three weeks for a cycle.
  BSA (body surface area) S-1 dosage <1.25 m2 80 mg/d
  * 1.25m2 - <1.5 m2 100 mg/d
  * 1.5 m2 120 mg/d
  Other Names: Tomudex, Gimeracil and oteracil porassium

SUMMARY:
The primary endpoint is to evaluate the Median disease progression free survival (mPFS).

DETAILED DESCRIPTION:
The primary endpoint is to evaluate the disease progression free survival (mPFS) of Raltitrexed combined with S-1 as treatment for patients with metastasizing colorectal cancer failed of standard chemotherapy

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Histologically or cytologically confirmed adenocarcinoma of the colon or rectum 3. No systemic chemotherapy for metastatic tumors

4. ECOG (Eastern Cooperative Oncology Group) 0-1 and expected survival period for 3 months or more 5. At least one measurable objective tumor lesions according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 6. ANC≥1.5*109/L；PLT≥80*109/L；HB≥90g/L；Total bilirubin ≤ 1.5 x the upper limit of normal (ULN) ; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x ULN (≤ 5 x ULN for subjects with liver involvement of their cancer)；ALB ≥ 30g/L; Serum creatinine ≤1.5(ULN) or glomerular filtration rate (GFR) ≥60 ml/min screening within 7 days 7. Progression during or within 3 months following the last administration of approved standard therapies which must include a fluoropyrimidine, oxaliplatin and irinotecan. Subjects treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy. Subjects who progress more than 6 months after completion of oxaliplatin containing adjuvant treatment must be retreated with oxaliplatin-based therapy to be eligible. Subjects who have withdrawn from standard treatment due to unacceptable toxicity warranting discontinuation of treatment and precluding retreatment with the same agent prior to progression of disease will also be allowed into the study. Subjects may have received prior treatment with Avastin (bevacizumab) and/or Erbitux (cetuximab)/Vectibix (panitumumab) (if KRAS WT) 8. Signed informed consent obtained before any study specific procedures. Subjects must be able to understand and willing to sign a written informed consent.

Exclusion Criteria:

1. Prior treatment with raltitrexed and gimeracil and oteracil potassium
2. Systemic anticancer therapy including cytotoxic therapy, signal transduction inhibitors, immunotherapy and hormonal therapy during this trial or within 4 weeks (or 6 weeks for mitomycin C) before starting to receive study medication.
3. Alcohol or drug addictions
4. Previous or concurrent cancer that is distinct in primary site or histology from colorectal cancer within 5 years prior to randomization EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)]
5. Any history of or currently known brain metastases
6. Multiple primary colorectal carcinoma
7. Concomitant participation or participation within the last 30 days in another clinical trial
8. There is an important organ failure or other serious diseases, including coronary artery disease, symptomatic cardiovascular disease or myocardial infarction within 12 months; serious neurological or psychiatric history; severe infection; actively disseminated vascula blood coagulation.
9. Extended field radiotherapy within 4 weeks or limited field radiotherapy within 2 weeks prior to randomization. Subjects must have recovered from all therapy-related toxicities. The site of previous radiotherapy should have evidence of progressive disease if this is the only site of disease.
10. Pregnant or breast-feeding subjects. Women of childbearing potential must have a pregnancy test performed a maximum of 7 days before start of treatment, and a negative result must be documented before start of treatment.
11. Pleural effusion or ascites that causes respiratory compromise (≥Common Terminology Criteria for Adverse Events [CTCAE]) Grade 2 dyspnea)
12. Subjects unable to swallow oral medications
13. Known history of human immunodeficiency virus (HIV) infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2015-12-25; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Median disease progression free survival (mPFS) of Raltitrexed combined with S-1 | at least 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Wei Jian Guo, doctor, Study Chair — Fudan University
Locations (1):
- Fudan University Cancer Hospital, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Huang M, Yang Y, Zhu X, Chen Z, Zhang W, Wang C, Zhang X, Qiu L, Zhang Z, Zhao X, Li W, Wang Y, Guo W. A prospective phase II study of raltitrexed combined with S-1 as salvage treatment for patients with refractory metastatic colorectal cancer. Asia Pac J Clin Oncol. 2021 Dec;17(6):513-521. doi: 10.1111/ajco.13511. Epub 2021 Feb 10. PMID 33567129